CLINICAL TRIAL: NCT05280717
Title: A Phase 1, Open-label, Randomized, Parallel Group, Single-dose Clinical Pharmacology Study to Investigate the Relative Bioavailability, Safety, and Tolerability of Two Different Concentrations of Sotrovimab Administered at Different Injection Sites, in Male or Female Healthy Participants Aged 18 to 65 Years
Brief Title: Relative Bioavailability, Safety, and Tolerability of Single-dose Sotrovimab Injection in Adults (COSMIC)
Acronym: COSMIC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part C cohort 1 was discontinued early in the context of evolving variants with increased fold changes in the in vitro half maximal inhibitory concentration (IC50) and uncertainty in the clinical relevance of these changes.
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-7831-5012; GSK Study 218128 (Other: GlaxoSmithKline)
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: COVID-19; Pharmacokinetics; Safety; Sotrovimab; Relative bioavailability; Healthy participants
MeSH Terms: conditions — COVID-19 | interventions — sotrovimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Treatment arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) (Experimental): Participants will receive a single 500 milligram (mg) of 62.5 milligram per milliliter (mg/mL) sotrovimab administered via two injections intramuscularly into the dorsogluteal muscle on Day 1.
  Interventions: Biological: sotrovimab
- Part A: Treatment arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) (Experimental): Participants will receive a single 500 mg of 100 mg/mL sotrovimab administered intramuscularly into the dorsogluteal muscle on Day 1.
  Interventions: Biological: sotrovimab
- Part A: Treatment arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) (Experimental): Participants will receive a single 500 mg of 100 mg/mL sotrovimab administered intramuscularly into the anterolateral thigh muscles on Day 1.
  Interventions: Biological: sotrovimab
- Part A: Treatment arm 4- Sotrovimab 100 mg/mL (Deltoid) (Experimental): Participants will receive a single 500 mg of 100 mg/mL sotrovimab administered two injections intramuscularly into the deltoid muscles on Day 1.
  Interventions: Biological: sotrovimab
- Part B: Sotrovimab (Experimental): Participants will receive 500 mg of 100 mg/mL and/or 62.5 mg/mL sotrovimab on Day 1.
  Interventions: Biological: sotrovimab
- Part C: Cohort 1-Sotrovimab (Experimental): Participants will receive a single 3000 mg of sotrovimab intravenous (IV) infusion over 60 minutes on Day 1.
  Interventions: Biological: sotrovimab
- Part C: Cohort 2-Sotrovimab (Experimental): Participants are planned to receive up to 3000 mg of sotrovimab intravenously on Day 1.
  Interventions: Biological: sotrovimab

INTERVENTIONS:
Biological: sotrovimab — via IM injection
  Arms: Part A: Treatment arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal)
Biological: sotrovimab — via IM injection
  Arms: Part A: Treatment arm 2- Sotrovimab 100 mg/mL (Dorsogluteal)
Biological: sotrovimab — via IM injection
  Arms: Part A: Treatment arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh)
Biological: sotrovimab — via IM injection
  Arms: Part A: Treatment arm 4- Sotrovimab 100 mg/mL (Deltoid)
Biological: sotrovimab — via IM injection
  Arms: Part B: Sotrovimab
Biological: sotrovimab — via IV injection
  Arms: Part C: Cohort 1-Sotrovimab
Biological: sotrovimab — via IV infusion
  Arms: Part C: Cohort 2-Sotrovimab

SUMMARY:
This clinical pharmacology study will evaluate the relative bioavailability, safety, and tolerability of two different concentrations of sotrovimab injections administered at different injection sites in male or female healthy participants aged 18 to 65 years. The study will be conducted in three parts (Part A, an optional Part B and Part C). Part B and Part C (cohort 2) were optional so they were not initiated. Part C cohort 1 was discontinued early in the context of evolving variants with increased fold changes in the in vitro half maximal inhibitory concentration (IC50) and uncertainty in the clinical relevance of these changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 18 to 65 years, inclusive.
* Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* For Part C, inclusion in the Japanese subgroup analysis, a participant must meet all of the following criteria: Japanese ancestry, defined as being a descendant of 4 ethnic Japanese grandparents and 2 ethnic Japanese parents.
* Body Mass Index (BMI) within the range of 18 to 30 kilogram per square meter (kg/m^2).
* Capable of giving signed informed consent

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Breast cancer within the past 10 years
* Abnormal blood pressure at Screening.
* Known hypersensitivity to any constituent present in the investigational product or history of severe hypersensitivity or anaphylaxis after receiving a COVID-19 vaccine
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Use of any over the counter or prescription medications unless permitted by the protocol or approved by the Investigator in conjunction with the GSK medical monitor.
* For Part A and Part B, any condition that would prohibit receipt of injections in the investigator's opinion, such as coagulation disorder, bleeding diathesis, or thrombocytopenia.
* Treatment with biologic agents (such as) within 3 months or 5 half-lives
* Receipt of convalescent plasma from a recovered COVID-19 participant or anti- severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) monoclonal antibody (mAb) within the last 3 months.
* Receipt of any vaccine within 48 hours prior to enrollment.
* Has received a SARS-CoV-2 vaccine but has not completed all doses in the series more than 28 days prior to Screening.
* Exposure to more than 4 new chemical entities (e.g., investigational pharmaceuticals) within 12 months prior to the first dosing day.
* Enrolment in any investigational vaccine study within the last 180 days or enrollment in any other investigational drug study within 30 days prior to Day 1 or within 5 half-lives
* Current enrolment or past participation in this clinical study.
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody test result at Screening or within 3 months prior to dosing.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* History of regular alcohol consumption within 6 months prior to the study.
* Regular use of known drugs of abuse.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Investigative Site, Riverside, California
  - Investigative Site, Atlantis, Florida
  - Investigative Site, Edgewater, Florida
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Binghamton, New York
  - Investigative Site, Yukon, Oklahoma
  - Investigative Site, Medford, Oregon
  - Investigative Site, Austin, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, West Jordan, Utah

REFERENCES:
- [Derived] Sanchez-Pearson Y, Moore J, Daniluk J, Bhangu S, Parra S, El Zailik A, Sarkar P, Aylott A, Moyo F, Peppercorn A, Skingsley A. Safety, Tolerability and Pharmacokinetics of a High-Dose, Rapid-Infusion Monoclonal Antibody: Phase I Results for Intravenous Sotrovimab 3000 mg. Drugs R D. 2025 Dec;25(4):367-376. doi: 10.1007/s40268-025-00530-9. Epub 2025 Dec 1. PMID 41324898
- [Derived] Moore J, Aylott A, Chen WH, Daniluk J, Hawes IA, Parra S, Sarkar P, Sanchez-Pearson Y, Turner M, Peppercorn A, Skingsley A. Safety and tolerability of intramuscular sotrovimab administered at different injection sites: results from the Phase 1 COSMIC study. MAbs. 2025 Dec;17(1):2456467. doi: 10.1080/19420862.2025.2456467. Epub 2025 Jan 29. PMID 39881564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3-part (Parts A, B and C) study. A total of 316 participants (216 participants in Part A and 100 participants in Part C) were enrolled in this study. Three participants were enrolled but not dosed. A total of 313 participants (215 in Part A and 98 in Part C) received Sotrovimab creating Safety Population (Safety Population consisted of all randomized participants who were exposed to study intervention).
Pre-assignment Details: Part B was optional and was not initiated in alignment with the strategic direction of the sotrovimab program and Part C Cohort-2 was optional and was not conducted as Part C Cohort-1 was stopped for programmatic reasons given the evolving Corona virus disease-19 (COVID-19) variant landscape. Hence, no participants were enrolled in Part B and Part C (Cohort-2) of the study.
Groups:
- Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal): Participants received a single 500 milligram (mg) of 62.5 milligram per milliliter (mg/mL) sotrovimab administered two injections intramuscularly into the dorsogluteal muscle on Day 1.
- Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal): Participants received a single 500 mg of 100 mg/mL sotrovimab administered intramuscularly into the dorsogluteal muscle on Day 1.
- Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh): Participants received a single 500 mg of 100 mg/mL sotrovimab administered intramuscularly into the anterolateral thigh muscles on Day 1.
- Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid): Participants received a single 500 mg of 100 mg/mL sotrovimab administered two injections intramuscularly into the deltoid muscles on Day 1.
- Part B: Sotrovimab: Participants were planned to receive 500 mg of 100 mg/mL and/or 62.5 mg/mL sotrovimab on Day 1.
- Part C: Cohort 1-Sotrovimab: Participants received a single 3000 mg of sotrovimab intravenous (IV) infusion over 60 minutes on Day 1.
- Part C: Cohort 2-Sotrovimab: Participants were planned to receive up to 3000 mg of sotrovimab intravenously on Day 1.
Period: Part A (Up to Week 35)
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) | Part B: Sotrovimab | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Started (Enrolled) | 72 | 72 | 36 | 36 | 0 | 0 | 0
Safety Population | 71 | 71 | 35 | 38 (Two participants randomized (one for treatment arm 2 and one for treatment arm 3), but dosed in treatment arm 4) | 0 | 0 | 0
Completed | 70 | 68 | 33 | 36 | 0 | 0 | 0
Not Completed | 2 | 4 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Randomized but not received treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant was randomized for treatment arm 2 but dosed in treatment arm 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant was randomized for treatment arm 3 but dosed in treatment arm 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part B (Up to Week 35)
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) | Part B: Sotrovimab | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (Up to Week 35)
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) | Part B: Sotrovimab | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Started (Enrolled) | 0 | 0 | 0 | 0 | 0 | 100 | 0
Safety Population | 0 | 0 | 0 | 0 | 0 | 98 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 96 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Enrolled but not received treatment | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Part B was not initiated in alignment with the strategic direction of the sotrovimab program and Part C Cohort-2 was not conducted as Part C Cohort-1 was stopped for programmatic reasons given the evolving Corona virus disease-19 (COVID-19) variant landscape. Hence, no participants were enrolled in Part B and Part C (Cohort-2). Baseline Characteristic data are reported for Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) | Part B: Sotrovimab | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab | Total
Number analyzed (Participants) | 71 | 71 | 35 | 38 | 0 | 98 | 0 | 313
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 |  | 2 |  | 2
  19-64 years | 70 | 71 | 35 | 38 |  | 96 |  | 310
  >=65 years | 1 | 0 | 0 | 0 |  | 0 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 21 | 20 |  | 47 |  | 169
  Male | 29 | 32 | 14 | 18 |  | 51 |  | 144
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 |  | 0 |  | 3
  Asian - Central/South Asian Heritage | 2 | 0 | 2 | 0 |  | 1 |  | 5
  Asian - East Asian Heritage | 0 | 0 | 0 | 1 |  | 2 |  | 3
  Asian - Japanese Heritage | 0 | 1 | 0 | 0 |  | 13 |  | 14
  Asian - South East Asian Heritage | 0 | 2 | 0 | 0 |  | 3 |  | 5
  Black or African American | 6 | 2 | 3 | 4 |  | 16 |  | 31
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 |  | 0 |  | 2
  White - Arabic/North African Heritage | 0 | 1 | 0 | 1 |  | 0 |  | 2
  White - White/Caucasian/European Heritage | 60 | 62 | 25 | 30 |  | 61 |  | 238
  Mixed Asian Race | 1 | 0 | 0 | 0 |  | 0 |  | 1
  Mixed Race | 2 | 0 | 1 | 0 |  | 1 |  | 4
  Missing | 0 | 1 | 2 | 1 |  | 1 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A (Treatment Arms 1 and 2): Area Under the Serum Concentration-time Curve (AUC) From Day 1 to Day 29 (AUC[D1 to 29]) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of sotrovimab. Pharmacokinetic (PK) parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: PK Population consisted of all participants in the Safety Population who had at least 1 non-missing PK assessment - i.e., PK sample collected and analyzed. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Geometric Mean (95% Confidence Interval); unit: Day*microgram per milliliter
Groups:
- Part A: Treatment Arm 1-Sotrovimab 62.5 mg/mL (Dorsogluteal): Participants received a single 500 milligram (mg) of 62.5 milligram per milliliter (mg/mL) sotrovimab administered two injections intramuscularly into the dorsogluteal muscle on Day 1.
- Part A: Treatment Arm 2-Sotrovimab 100 mg/mL (Dorsogluteal): Participants received a single 500 mg of 100 mg/mL sotrovimab administered intramuscularly into the dorsogluteal muscle on Day 1.
Arm/Group | Part A: Treatment Arm 1-Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2-Sotrovimab 100 mg/mL (Dorsogluteal)
Number analyzed (Participants) | 65 | 68
Day*microgram per milliliter | 944.94 [844.74 to 1057.02] | 950.67 [837.05 to 1079.72]
Statistical Analysis 1: Comparison: Part A: Treatment Arm 1-Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 2-Sotrovimab 100 mg/mL (Dorsogluteal); Test type: Other; Ratio of geometric least square mean = 0.9821, 90% CI 2-sided [0.8825 to 1.0930] — The ratio estimate and 90% confidence interval were obtained from an Analysis of covariance (ANCOVA) model, with AUC(D1- 29) as the dependent variable, and sex, baseline body mass index and treatment as covariates

2. Primary Outcome: Part A (Treatment Arms 1 and 2): Maximum Observed Concentration (Cmax) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of sotrovimab. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: PK Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | Part A: Treatment Arm 1-Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2-Sotrovimab 100 mg/mL (Dorsogluteal)
Number analyzed (Participants) | 71 | 70
Microgram per milliliter | 37.91 [33.76 to 42.57] | 44.10 [39.23 to 49.57]
Statistical Analysis 1: Comparison: Part A: Treatment Arm 1-Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 2-Sotrovimab 100 mg/mL (Dorsogluteal); Test type: Other; Ratio of geometric least square mean = 1.1258, 90% CI 2-sided [1.0108 to 1.2539] — The ratio estimate and 90% confidence interval were obtained from an ANCOVA model, with Cmax as the dependent variable, and sex, baseline body mass index and treatment as covariates

3. Primary Outcome: Part A (Treatment Arms 1 and 2): Number of Participants With Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESI) and Common (>=5%) Non-serious Adverse Events (Non-SAEs) Through Day 29
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life- threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before. Adverse events which were not Serious were considered as non-serious adverse events. Number of participants who had common (>=5%) non-SAEs and SAEs are presented. AESIs included hypersensitivity reactions and injection site reactions based on a predefined list of terms.
Time Frame: Up to Day 29
Population: Safety Population consisted of all randomized participants who were exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment Arm 1-Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2-Sotrovimab 100 mg/mL (Dorsogluteal)
Number analyzed (Participants) | 71 | 71
Participants
  Non-SAEs | 27 | 20
  SAEs | 0 | 0
  AESIs | 24 | 15

4. Primary Outcome: Part C (Cohorts 1 and 2): Number of Participants With SAEs, AESIs and Common (>=5%) Non-SAEs Through Day 29
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before. Adverse events which were not Serious were considered as non-serious adverse events. Number of participants who had common (>=5%) non-SAEs and SAEs are presented. AESI included hypersensitivity reaction based on a predefined list of terms.
Time Frame: Up to Day 29
Population: Safety Population. Data was not collected as no participants were enrolled in Part C: Cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Number analyzed (Participants) | 98 | 0
Participants
  Non-SAEs | 9 |
  SAEs | 0 |
  AESIs | 1 |

5. Secondary Outcome: Part A (Treatment Arms 1, 3 and 4): AUC(D1 to 29) Following Administration of Sotrovimab
Description: as for outcome 2
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Day*microgram per milliliter
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid)
Number analyzed (Participants) | 65 | 31 | 37
Day*microgram per milliliter | 944.94 [844.74 to 1057.02] | 1849.83 [1691.90 to 2022.50] | 1525.17 [1424.83 to 1632.58]
Statistical Analysis 1: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh); Test type: Other; Ratio of geometric least square mean = 1.8760, 90% CI 2-sided [1.6391 to 2.1472] — The ratio estimate and 90% confidence interval were obtained from an ANCOVA model, with AUC(D1-29) as the dependent variable, and sex, baseline body mass index and treatment as covariates
Statistical Analysis 2: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid); Test type: Other; Ratio of geometric least square mean = 1.5991, 90% CI 2-sided [1.4086 to 1.8153] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Part A (Treatment Arms 1, 3 and 4): Cmax Following Administration of Sotrovimab
Description: as for outcome 2
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid)
Number analyzed (Participants) | 71 | 35 | 38
Microgram per milliliter | 37.91 [33.76 to 42.57] | 82.08 [75.75 to 88.93] | 64.99 [60.50 to 69.82]
Statistical Analysis 1: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh); Test type: Other; Ratio of geometric least square mean = 2.0798, 90% CI 2-sided [1.8223 to 2.3737] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid); Test type: Other; Ratio of geometric least square mean = 1.6955, 90% CI 2-sided [1.4913 to 1.9276] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Part B: AUC(D1-29) Following Administration of Sotrovimab
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of sotrovimab.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Sotrovimab
Number analyzed (Participants) | 0

8. Secondary Outcome: Part B: Cmax Following Administration of Sotrovimab
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of sotrovimab.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Sotrovimab
Number analyzed (Participants) | 0

9. Secondary Outcome: Part C (Cohorts 1 and 2): AUC(D1-29) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of sotrovimab in Cohort 1. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1: Pre-dose, end of infusion, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: PK Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. Data was not collected as no participants were enrolled in Part C: Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Number analyzed (Participants) | 82 | 0
Day*microgram per milliliter | 12064.44 (21.50) |

10. Secondary Outcome: Part C (Cohorts 1 and 2): Cmax Following Administration of Sotrovimab
Description: as for outcome 9
Time Frame: Day 1: Pre-dose, end of infusion, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15 and 29 post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Number analyzed (Participants) | 86 | 0
Microgram per milliliter | 1124.32 (21.69) |

11. Secondary Outcome: Part A (Treatment Arms 1, 2, 3 and 4): Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUCinf) Following Administration of Sotrovimab at 3 Injection Sites
Description: as for outcome 2
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 140, 168 (Week 24) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid)
Number analyzed (Participants) | 49 | 59 | 32 | 34
Day*microgram per milliliter | 3979.55 (39.88) | 3851.37 (47.68) | 6397.59 (20.17) | 5511.58 (26.28)
Statistical Analysis 1: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal); Test type: Other; Ratio of geometric least square mean = 0.9476, 90% CI 2-sided [0.8578 to 1.0469] — The ratio estimate and 90% confidence interval were obtained from an ANCOVA model, with AUCinf as the dependent variable, and sex, baseline body mass index and treatment as covariates
Statistical Analysis 2: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh); Test type: Other; Ratio of geometric least square mean = 1.5482, 90% CI 2-sided [1.3770 to 1.7407] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) vs Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid); Test type: Other; Ratio of geometric least square mean = 1.4167, 90% CI 2-sided [1.2627 to 1.5894] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Part B: AUCinf Following Administration of Sotrovimab at up to 2 Injection Sites
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of sotrovimab.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 140, 168 (Week 24) post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Sotrovimab
Number analyzed (Participants) | 0

13. Secondary Outcome: Part A (Treatment Arms 1, 2, 3 and 4): Serum Concentration Following Administration of Sotrovimab
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of sotrovimab.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 140, 168 post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid)
Number analyzed (Participants) | 71 | 70 | 35 | 38
Microgram per milliliter
  Day 1: Pre-dose: number analyzed (Participants) | 71 | 69 | 34 | 38
  Day 1: Pre-dose | 0.0 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 0.0 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 0.0 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 0.0 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed).
  Day 1: 1 hour: number analyzed (Participants) | 61 | 60 | 27 | 38
  Day 1: 1 hour | 0.6 (0.97) | 1.6 (8.03) | 5.0 (14.58) | 1.4 (1.53)
  Day 1: 2 hours: number analyzed (Participants) | 71 | 69 | 35 | 37
  Day 1: 2 hours | 1.8 (3.29) | 1.3 (1.39) | 4.8 (13.05) | 3.1 (2.10)
  Day 1: 6 hours: number analyzed (Participants) | 70 | 70 | 35 | 38
  Day 1: 6 hours | 6.7 (7.17) | 11.0 (15.56) | 14.1 (15.10) | 12.7 (7.00)
  Day 1: 8 hours | 9.9 (10.46) | 11.1 (10.93) | 21.2 (17.85) | 18.2 (12.51)
  Day 2 | 19.9 (14.34) | 21.7 (15.61) | 45.1 (24.51) | 38.9 (16.96)
  Day 3 | 30.0 (18.26) | 34.4 (21.40) | 68.8 (22.74) | 53.5 (17.60)
  Day 5: number analyzed (Participants) | 71 | 70 | 34 | 38
  Day 5 | 36.2 (18.95) | 41.8 (22.03) | 80.3 (15.63) | 63.3 (14.41)
  Day 8: number analyzed (Participants) | 70 | 70 | 35 | 38
  Day 8 | 38.2 (17.92) | 42.5 (20.95) | 78.9 (14.65) | 62.6 (13.77)
  Day 15: number analyzed (Participants) | 70 | 70 | 33 | 38
  Day 15 | 38.4 (16.78) | 41.6 (17.43) | 67.8 (17.61) | 57.7 (11.60)
  Day 29: number analyzed (Participants) | 70 | 69 | 33 | 38
  Day 29 | 34.3 (12.48) | 35.5 (14.13) | 59.5 (12.24) | 49.9 (13.02)
  Day 57: number analyzed (Participants) | 71 | 69 | 33 | 38
  Day 57 | 24.5 (8.71) | 24.9 (10.91) | 39.3 (11.65) | 33.2 (8.36)
  Day 85: number analyzed (Participants) | 70 | 68 | 33 | 38
  Day 85 | 17.6 (5.74) | 17.5 (7.51) | 27.3 (7.73) | 25.8 (10.53)
  Day 140: number analyzed (Participants) | 70 | 68 | 33 | 38
  Day 140 | 9.7 (3.84) | 10.1 (8.66) | 14.6 (4.53) | 13.0 (3.83)
  Day 168: number analyzed (Participants) | 69 | 68 | 33 | 38
  Day 168 | 7.6 (3.46) | 6.9 (3.09) | 10.1 (2.73) | 10.3 (4.01)

14. Secondary Outcome: Part B: Serum Concentration Following Administration of Sotrovimab
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic analysis of sotrovimab.
Time Frame: Day 1: Pre-dose, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 140, 168 post-dose
Population: PK Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Sotrovimab
Number analyzed (Participants) | 0

15. Secondary Outcome: Part C: Serum Concentration Following Administration of Sotrovimab
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of sotrovimab in Cohort 1.
Time Frame: Day 1: Pre-dose, end of infusion, 1, 2, 6 and 8 hours post-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 140, 168 post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Number analyzed (Participants) | 98 | 0
Microgram per milliliter
  Day 1: Pre-dose: number analyzed (Participants) | 87 | 0
  Day 1: Pre-dose | 0.0 (NA) — Standard deviation could not be calculated due to high proportion of NQ values (>30% of values were imputed). |
  Day 1: End of infusion: number analyzed (Participants) | 87 | 0
  Day 1: End of infusion | 1069.2 (261.39) |
  Day 1: 1 hour | 976.3 (265.40) |
  Day 1: 2 hours | 993.3 (241.85) |
  Day 1: 6 hours | 921.5 (235.27) |
  Day 1: 8 hours | 934.3 (224.54) |
  Day 2: number analyzed (Participants) | 96 | 0
  Day 2 | 802.9 (193.80) |
  Day 3: number analyzed (Participants) | 97 | 0
  Day 3 | 685.1 (168.11) |
  Day 5 | 584.8 (149.55) |
  Day 8 | 470.9 (110.32) |
  Day 15: number analyzed (Participants) | 97 | 0
  Day 15 | 407.4 (104.25) |
  Day 29 | 320.2 (74.93) |
  Day 57: number analyzed (Participants) | 85 | 0
  Day 57 | 223.9 (71.55) |
  Day 85: number analyzed (Participants) | 85 | 0
  Day 85 | 159.1 (56.97) |
  Day 140: number analyzed (Participants) | 95 | 0
  Day 140 | 85.9 (32.60) |
  Day 168: number analyzed (Participants) | 96 | 0
  Day 168 | 61.0 (30.72) |

16. Secondary Outcome: Part A (Treatment Arms 1, 2, 3 and 4): Number of Participants With SAEs, AESI and Common (>=5%) Non-SAEs Through Day 29 and Week 35
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before. Adverse events which were not Serious were considered as non-serious adverse events. Number of participants who had common (>=5%) non-SAEs and SAEs are presented. AESIs included hypersensitivity reactions and injection site reactions based on a predefined list of terms.
Time Frame: Up to Day 29 and Up to Week 35
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid)
Number analyzed (Participants) | 71 | 71 | 35 | 38
Participants
  Up to Day 29: SAEs | 0 | 0 | 0 | 0
  Up to Day 29: Non-SAEs | 27 | 20 | 13 | 20
  Up to Day 29: AESIs | 24 | 15 | 13 | 18
  Up to Week 35: SAEs | 1 | 1 | 0 | 0
  Up to Week 35: Non-SAEs | 29 | 22 | 13 | 20
  Up to Week 35: AESIs | 25 | 15 | 13 | 18

17. Secondary Outcome: Part B: Number of Participants With SAEs, AESIs and Common (>=5%) Non-SAEs Through Day 29 and Week 35
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before. AESIs included hypersensitivity reactions and injection site reactions based on a predefined list of terms.
Time Frame: Up to Day 29 and Up to Week 35
Population: Safety Population. Data was not collected as no participants were enrolled in Part B.
Arm/Group | Part B: Sotrovimab
Number analyzed (Participants) | 0

18. Secondary Outcome: Part C: Number of Participants With SAEs, AESIs and Common (>=5%) Non-SAEs Through Week 35
Description: as for outcome 16
Time Frame: Up to Week 35
Population: Safety Population. Data was not collected as no participants were enrolled in Part C: Cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
Number analyzed (Participants) | 98 | 0
Participants
  SAEs | 0 |
  Non-SAEs | 9 |
  AESIs | 2 |

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-SAEs were collected up to Week 35 in Part A and Part C (Cohort-1) of the study
Description: Safety Population. All-cause mortality, non-SAEs and SAEs were not collected in Part B and Part C (Cohort-2) as no participants were enrolled. Data is presented for Part A and Part C (Cohort-1) only as data was not collected in Part B and Part C (Cohort-2) due to study stopped and Part B and Part C (Cohort-2) were not initiated.
Arm/Group | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) | Part B: Sotrovimab | Part C: Cohort 1-Sotrovimab | Part C: Cohort 2-Sotrovimab
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/71 | 0/35 | 0/38 | 0/0 | 0/98 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/71 | 1/71 | 0/35 | 0/38 | 0/0 | 0/98 | 0/0
Other Adverse Events (participants affected / at risk) | 29/71 | 22/71 | 13/35 | 20/38 | 0/0 | 9/98 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) (N=71) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) (N=71) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) (N=35) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) (N=38) | Part B: Sotrovimab (N=0) | Part C: Cohort 1-Sotrovimab (N=98) | Part C: Cohort 2-Sotrovimab (N=0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment Arm 1- Sotrovimab 62.5 mg/mL (Dorsogluteal) (N=71) | Part A: Treatment Arm 2- Sotrovimab 100 mg/mL (Dorsogluteal) (N=71) | Part A: Treatment Arm 3- Sotrovimab 100 mg/mL (Anterolateral Thigh) (N=35) | Part A: Treatment Arm 4- Sotrovimab 100 mg/mL (Deltoid) (N=38) | Part B: Sotrovimab (N=0) | Part C: Cohort 1-Sotrovimab (N=98) | Part C: Cohort 2-Sotrovimab (N=0)
Injection site pain (General disorders) | 25 | 14 | 9 | 18 | 0 | 0 | 0
Injection site induration (General disorders) | 2 | 2 | 4 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 7 | 4 | 0 | 4 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 9 | 0
Headache (Nervous system disorders) | 1 | 6 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT05280717/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT05280717/SAP_001.pdf